CLINICAL TRIAL: NCT07029815
Title: Assessment of Er:YAG (Yttrium-aluminium-garnet) Laser-Assisted Surgical Treatment in Medication-Related Osteonecrosis of the Jaw (MRONJ): A Clinical Trial
Brief Title: Assessment of Er:YAG Laser-Assisted Surgical Treatment in Medication-Related Osteonecrosis of the Jaw (MRONJ): A Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KB-27/2021
Record Dates: First submitted 2025-06-02; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-05

CONDITIONS: Medication-Related Osteonecrosis of Jaw
MeSH Terms: interventions — Radiation; Lasers, Solid-State

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients treated with the Er:YAG laser (Experimental)
  Interventions: Procedure: irradiation with Er:YAG laser
- Patients treated with the conventional surgery (Active Comparator)
  Interventions: Procedure: Tissue preparation

INTERVENTIONS:
Procedure: irradiation with Er:YAG laser — An Er:YAG laser (LightTouch, LightInstruments, Yokneam, Israel) was used with the following parameters: 400mJ (millijoules), 6W (Watt), 15Hz (Hertz), 5/8 water cooling, laser tip with a diameter of 800 microns. Tissue debridement continued until hard, healthy, lively bleeding bone was exposed, indicative of normal bone.
  Arms: Patients treated with the Er:YAG laser
Procedure: Tissue preparation — Rose-shaped rotary drills (8 mm diameter) were used with water cooling at a speed not exceeding 40.000 rpm. Tissue preparation limits were consistent with those used for the Er:YAG laser group.
  Arms: Patients treated with the conventional surgery

SUMMARY:
The aim of this study is assessing the effectiveness of the Er:YAG laser in relation to the use of conventional surgery in the treatment of drug-induced osteonecrosis of the jaws (MRONJ). The study compares two main treatments for advanced cases of MRONJ or cases that do not show improvement despite conservative or non-surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of MRONJ

Exclusion Criteria:

* head and neck radiotherapy
* cases requiring hospital admission due to poor general condition

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Complications | Up to 6 months
  Occurrence or absence of complications

OTHER OUTCOMES:
Severity of Osteonecrosis | 3 and 6 months after treatment.
  Incidence of grade II/III necrosis or no severe necrosis

CONTACTS AND LOCATIONS:
Overall Officials: Kinga Grzech-Leśniak, DDS, MS PhD, Study Director — Dental Surgery Department, Wroclaw Medical University, Krakowska st. 26, 50-425 Wroclaw, Poland and Department of Periodontics, School of Dentistry Virginia Commonwealth University, 12th St, Richmond, VA 23298, USA; Marzena Dominiak, Prof. dr hab n. med., Study Chair — Dental Surgery Department, Wroclaw Medical University, Krakowska st. 26, 50-425 Wroclaw, Poland
Locations (1):
- Wroclaw Medical University, Wroclaw, Poland

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/15/NCT07029815/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/15/NCT07029815/ICF_001.pdf